CLINICAL TRIAL: NCT06875375
Title: A Clinical Study on the Safety and Efficacy of Probiotic LH76 in Modulating Gut Microbiota and Enhancing Intestinal Health in Healthy Adults
Brief Title: The Role of Probiotic LH76 in Human Gut Health
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WK20250309
Record Dates: First submitted 2025-03-08; First posted 2025-03-13 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Gut Microbiota Modulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Probiotic group (Experimental)
  Interventions: Dietary Supplement: probiotic LH76

INTERVENTIONS:
Dietary Supplement: probiotic LH76 — Intervention with LH76 (30 billion CFU/ day, 3g) was administered daily for 8 weeks. Store in a cool, dry place.
  Arms: Probiotic group
Dietary Supplement: Placebo — Every day to give 3 g maltodextrin intervention for 8 weeks. Store in a cool and dry place.
  Arms: Placebo group

SUMMARY:
This study aims to evaluate the safety and efficacy of the probiotic LH76 as a dietary supplement in healthy adults. The research will assess its effects on gut microbiota composition, intestinal health, and immune function compared to a placebo. Key outcomes include changes in microbial diversity, intestinal barrier integrity, and immune response markers over the intervention period. The findings will contribute to understanding the potential health benefits of LH76 and its role in supporting gut and immune health.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to undergo 3 follow-up visits during the intervention period Be willing to provide blood, urine and stool samples 2 times during the intervention period
2. Willing to self-administer probiotic or placebo once a day during the intervention period
3. Good eyesight, can read and write, can wear glasses
4. Have good hearing and be able to hear and understand all instructions during the intervention

Exclusion Criteria:

1. Digestive diseases, mainly gastrointestinal diseases (celiac disease, ulcerative colitis, Crohn's disease)
2. Have a serious neurological condition (epilepsy, stroke, severe head trauma, meningitis in the last 10 years, brain surgery, brain tumor, prolonged coma - not including general anaesthesia)
3. Have received/are receiving treatment for the following mental disorders: alcohol/drug/substance abuse dependence, schizophrenia, psychosis, bipolar disorder
4. Take medication for depression or low mood Internal organ failure (heart, liver or kidney failure, etc.)
5. Have received radiation or chemotherapy in the past
6. Have undergone a general anesthesia procedure/procedure within the past three years, or plan to undergo a general anesthesia procedure/procedure within the next 3 months during this trial period
7. Have had hepatitis (hepatitis B, hepatitis C), HIV or syphilis in the past Open Contacts/Locations

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-11 (Estimated); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-10-26 (Estimated)

PRIMARY OUTCOMES:
Changes in Gut Microbiota Composition in Response to LH76 Supplementation | Week 0 and Week 8
  This study assesses the impact of LH76 supplementation on gut microbiota diversity and composition using high-throughput sequencing. The primary objective is to determine whether LH76 supplementation leads to significant improvements in gut microbiota balance compared to a placebo. Changes in microbial diversity, relative abundance of beneficial bacteria will be analyzed to assess the probiotic's effectiveness.